CLINICAL TRIAL: NCT02030509
Title: Quick Diagnostic Program for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Rosa Rosell Ferrer, PhD MD, Corporacion Parc Tauli
Other Study IDs: CSPT_ORL_2014_1
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Cancer of Head and Neck
Keywords: cancer diagnosis
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- New diagnosed patients of head and neck cancer: New diagnosed patients of head and neck cancer
  Interventions: Other: Quick diagnosis program
- Old diagnosed head and neck cancer patients

INTERVENTIONS:
Other: Quick diagnosis program
  Groups: New diagnosed patients of head and neck cancer

SUMMARY:
Head and neck cancer would be suitable for quick diagnostic programs because their initial symptoms are easy detectable and the curation rates in the initial stages are very high.

Actually the stages at diagnosis are about 30% in initial stages and 70% in advanced stages.

The hypothesis of this study is that a program for quick referral of patients with symptoms of head and neck cancer would help early diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms of head and neck cancer in the Hospital reference area

Exclusion Criteria:

* Patients already diagnosed when refered to Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with symptoms of head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Time from symptom onset to diagnosis | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona, Spain